CLINICAL TRIAL: NCT05077423
Title: A Phase 1, Open-label, Dose-escalation Trial of CD33xCD3 Bispecific Antibody in Pediatric Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: A Phase 1 Trial of CD33xCD3 BsAb in Pediatric Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to business priorities
Sponsor: Y-mAbs Therapeutics (Industry)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 801
Record Dates: First submitted 2021-09-30; First posted 2021-10-14 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-11

CONDITIONS: AML, Childhood
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: open-label, single-arm, dose-escalation consisting of up to 12 cycles
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subcutaneous administration of CD33*CD3 BsAb up to 12 cycles (Experimental): Subcutaneous administration of CD33*CD3 BsAb up to 12 cycles
  Interventions: Drug: CD33*CD3 BsAb

INTERVENTIONS:
Drug: CD33*CD3 BsAb — CD33xCD3 is a bispecific monoclonal antibody, which specifically targets CD33 on the AML blasts and CD3 on the T cells
  Other Names: CD33xCD3

SUMMARY:
Pediatric patients (<21 years at study entry) with relapsed or refractory acute myeloid leukemia (AML) will be treated with CD33*CD3 a bispecific antibody to investigate the safety and tolerability of the drug.

DETAILED DESCRIPTION:
This is an open label, first in human dose escalation trial in pediatric patients with relapsed or refractory acute myeloid leukemia to assess the safety and tolerability of increasing doses of CD33xCD3 BsAb administered subcutaneously.

A modified Bayesian Optimal Interval Design (mBOIN) design will be applied. The trial will start with accelerated titration using single patient cohorts until one grade ≥2 AE not clearly associated to underlying disease, thereafter the trial will continue with mBOIN titration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from legal guardian(s), patient and/or child obtained in accordance with local regulations. Pediatric patients must provide assent as required by local regulations
* Age ≥2 years, and ≤21 years, and a minimum body weight of ≥11 kg
* Histologically confirmed relapsed or refractory AML (except acute promyelocytic leukemia) with no therapeutic options that may provide clinical benefit. Disease burden ≥5.0% in the bone marrow meets definition for enrollment.
* Karnofsky performance status ≥50 for ≥16 years / Lansky performance status ≥50 for <16 years
* White blood cells (WBC) ≤25 x 109/L (may receive hydroxyurea to bring WBC count down prior to first dose of CD33xCD3 BsAb and during Cycle 1 or low dose cytarabine up to 48 h prior to first dose of CD33xCD3 BsAb)
* Central Nervous System (CNS) disease as per Children's Oncology Group

  * Patients must have the status of CNS1 and no clinical signs or neurologic symptoms suggestive of CNS leukemia, such as cranial palsy
  * Patients with CNS3 or CNS2 status may receive antecedent intrathecal chemotherapy to achieve CNS1 status prior to trial entry
  * Patients with a history of CNS chloromatous disease are required to have no radiographic evidence of disease prior to enrollment
* Has acceptable liver and kidney laboratory values
* Patient must have recovered from acute toxic effects of prior anti-cancer therapies prior to first dose of CD33xCD3 BsAb

Exclusion Criteria:

* History of uncontrolled seizure. If on anti-convulsant and/or seizures are well controlled as per treating physician enrollment is acceptable
* Acute promyelocytic leukemia with PML-RARA genetic abnormality according to WHO classification or t(15;17)
* Isolated extramedullary AML
* Clinically significant graft-versus-host disease (GvHD) secondary to prior allogeneic transplantation. No immunosuppressive therapy for ≥14 days prior to first dose, except for topical corticosteroids for minor rash (<5% of BSA) or adrenal replacement therapy
* Patient known to have one of the following genetic syndromes: Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Nijmegen breakage syndrome, Kostmann syndrome, Shwachman Diamond syndrome or any known bone marrow failure syndrome where increased risk for toxicity may be expected as judged by the Investigator
* Treatment with another investigational agent under the following conditions:

  * Within two weeks (four weeks for biologics) before first administration of CD33xCD3 BsAb; or
  * Patient has persistent toxicities from prior anti-leukemic therapies which are determined to be relevant by the Investigator

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities (DLTs) | 28 days
  Occurrence of DLTs during a DLT period .
Occurrence of Adverse Events | 52 weeks
  Occurrence of Adverse Events during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Pollard, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (13):
- United States (13):
  - Children's of Alabama/University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Riley Hospital for Children - Indiana University, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No